CLINICAL TRIAL: NCT07205263
Title: A Multicenter, Randomized, Controlled, Umbrella Trial for Minimally Invasive Neurosurgery With Al-assisted Robotic Guidance for Hemorrhagic Stroke (RAINBOW-ICH)
Brief Title: RAINBOW-ICH Trial of AI Guided Minimally Invasive Neurosurgery for ICH
Acronym: RAINBOW-ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Huashan Hospital (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023ZD0505000
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-08

CONDITIONS: Basal Ganglia Hemorrhage; Intraventricular Hemorrhage; Brainstem Stroke; Intracranial Hemorrhage, Spontaneous
Keywords: Umbrella Trial; Intraventricular hemorrhage; Brainstem Stroke; Robotic-guided; Basal Ganglia Hemorrhage; Minimally invasive surgery
MeSH Terms: conditions — Basal Ganglia Hemorrhage; Brain Stem Infarctions; Intracranial Hemorrhages

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAINBOW-LBH substudy (Experimental): This substudy is a prospective, multicenter, randomized, controlled, parallel-group trial with blinded endpoint assessment to evaluate the efficacy and safety of AI-assisted robotic-guided endoscopic hematoma evacuation for patients with large basal ganglia hemorrhage (LBH).
  Interventions: Procedure: AI-assisted robotic-guided endoscopic hematoma evacuation; Procedure: Conventional craniotomy
- RAINBOW-MBH substudy (Experimental): This substudy is a prospective, multicenter, randomized, controlled, parallel-group trial with blinded endpoint assessment to evaluate AI-assisted robotic-guided puncture and hematoma evacuation for patients with moderate basal ganglia hemorrhage (MBH).
  Interventions: Procedure: AI-assisted robotic-guided puncture and hematoma evacuation; Other: Standard medical management
- RAINBOW-IVH substudy (Experimental): This substudy is a prospective, multicenter, randomized, controlled, parallel-group trial with blinded endpoint assessment to evaluate AI-assisted robotic-guided endoscopic ventricular hematoma evacuation with external ventricular drainage for patients with intraventricular hemorrhage (IVH)
  Interventions: Procedure: AI-assisted robotic-guided endoscopic ventricular hematoma evacuation plus external ventricular drainage; Procedure: External ventricular drainage (EVD)
- RAINBOW-BSH substudy (Experimental): This substudy is a prospective, multicenter, randomized, controlled, parallel-group trial with blinded endpoint assessment to evaluate AI-assisted robotic-guided puncture and hematoma evacuation for patients with brainstem hemorrhage (BSH).
  Interventions: Procedure: AI-assisted robotic-guided puncture and hematoma evacuation; Other: Standard medical management

INTERVENTIONS:
Procedure: AI-assisted robotic-guided endoscopic hematoma evacuation — Surgical removal of hematoma using AI-assisted robotic-guided stereotactic navigation and endoscopic aspiration techniques.
  Arms: RAINBOW-LBH substudy
Procedure: Conventional craniotomy — Standard open surgical evacuation of hematoma through craniotomy.
  Arms: RAINBOW-LBH substudy
Procedure: AI-assisted robotic-guided puncture and hematoma evacuation — AI-assisted robotic-guided stereotactic puncture and aspiration of hematoma.
  Arms: RAINBOW-BSH substudy; RAINBOW-MBH substudy
Other: Standard medical management — Guideline-based conservative therapy without surgical hematoma evacuation.
  Arms: RAINBOW-BSH substudy; RAINBOW-MBH substudy
Procedure: AI-assisted robotic-guided endoscopic ventricular hematoma evacuation plus external ventricular drainage — AI-assisted robotic-guided endoscopic evacuation of ventricular hematoma combined with external ventricular drainage.
  Arms: RAINBOW-IVH substudy
Procedure: External ventricular drainage (EVD) — Conventional ventricular catheter placement for hematoma drainage.
  Arms: RAINBOW-IVH substudy

SUMMARY:
Intracerebral hemorrhage (ICH) is one of the most devastating forms of stroke, with high rates of death and disability worldwide. Despite advances in medical and surgical care, effective therapeutic options remain limited. To address this gap, the RAINBOW-ICH trial has been designed as a nationwide, multicenter, randomized umbrella trial evaluating the efficacy and safety of AI-assisted, robotic-guided minimally invasive neurosurgery compared with conventional strategies across major ICH subtypes.

Under a single master protocol, RAINBOW-ICH incorporates multiple parallel randomized controlled substudies, each targeting a distinct ICH population-large basal ganglia hemorrhage, moderate basal ganglia hemorrhage, intraventricular hemorrhage, and brainstem hemorrhage. This umbrella design allows efficient use of resources while generating high-quality evidence tailored to the specific needs of different ICH subgroups, thereby supporting a more patient-centered approach to care.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is a leading cause of stroke-related mortality and long-term disability worldwide. Conventional surgical techniques, including craniotomy and catheter-based drainage, are often associated with significant procedural risks and variable outcomes across clinical settings. Minimally invasive approaches have been proposed to reduce surgical trauma, improve precision, and enhance recovery. Recent studies, such as the ENRICH trial, have provided encouraging evidence that selected patients may benefit from early minimally invasive hematoma evacuation, though results remain heterogeneous and further validation is needed across different ICH subtypes and populations.

The RAINBOW-ICH trial has been established to address this critical gap by systematically evaluating the role of AI-assisted, robotic-guided minimally invasive neurosurgery. Advances in robotics and artificial intelligence have enabled neurosurgeons to achieve greater precision in hematoma evacuation, minimize surgical injury, and improve reproducibility of complex procedures. RAINBOW-ICH is designed as a nationwide, multicenter umbrella trial, conducted under a single master protocol, with multiple parallel randomized controlled substudies. Each substudy focuses on a distinct ICH population and directly compares AI-assisted robotic-guided hematoma evacuation with the conventional standard of care relevant to that subgroup. Specifically, RAINBOW-LBH (NCT06484374) evaluates patients with large basal ganglia hemorrhage, RAINBOW-MBH (NCT06465719) addresses moderate basal ganglia hemorrhage, RAINBOW-IVH (NCT06486480) investigates intraventricular hemorrhage, and RAINBOW-BSH (NCT06459427) targets brainstem hemorrhage.

Within each substudy, participants are randomized to receive either AI-assisted robotic-guided minimally invasive neurosurgery or the control intervention, such as conventional craniotomy, external ventricular drainage, or optimized medical management. All substudies are conducted as multicenter RCTs across China, ensuring adequate and rapid recruitment, generalizability, and rigorous evaluation of interventions in diverse clinical environments.

By integrating minimally invasive neurosurgical technologies with a unified multicenter umbrella trial design, RAINBOW-ICH represents the first large-scale effort in China to rigorously test and compare surgical strategies for ICH. The findings are expected to generate high-quality evidence, refine clinical practice, and ultimately improve neurological outcomes for patients with this devastating disease.

ELIGIBILITY:
Umbrella Trial Inclusion Criteria:

1. Age ≥18 years；
2. Clinical diagnosis of spontaneous hemorrhagic stroke；

Umbrella Trial Exclusion Criteria:

1. Radiologically diagnosed cerebrovascular abnormalities, as well as ischemic infarction converting to intracerebral hemorrhage, or recent (within 1 year) recurrence of intracerebral hemorrhage；

Each substudy will specify additional inclusion and exclusion criteria in the respective Substudy-specific Registration. Patients who fulfill the overall umbrella trial criteria will be assessed for enrollment into each substudy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Utility-weighted modified Rankin Scale (UW-mRS) | Umbrella level time frame: 6 months; Substudy specific time frame may differ (details will be included in substudy-specific registration)
  The mRS is a 7-level ordinal scale used to evaluate functional outcomes after stroke. The categories are defined as follows:
  0 = No symptoms
  1. = No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. = Moderate disability. Requires some help, but able to walk unassisted.
  4. = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. = Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. = Dead Utility-weighted modified Rankin Scale (UW-mRS) , which applies utility values to each mRS category as shown below： mRS 0= UW-mRS 1；mRS 1= UW-mRS 0.91; mRS 2= UW-mRS 0.76; mRS 3= UW-mRS 0.65; mRS 4= UW-mRS 0.33; mRS 5= UW-mRS 0; mRS 6= UW-mRS 0.

SECONDARY OUTCOMES:
Ordinal shift in modified Rankin Scale | Umbrella level time frame: 6 months; Substudy specific time frame may differ (details will be included in substudy-specific registration)
  Ordinal shift analysis of the modified Rankin Scale (mRS), which measures the degree of disability or dependence in daily activities after stroke. The scale ranges from 0 (no symptoms) to 6 (death). This outcome assesses whether there is a shift toward better or worse functional status across the full ordinal distribution of mRS scores.
Excellent functional neurological outcome | Umbrella level time frame: 6 months; Substudy specific time frame may differ (details will be included in substudy-specific registration)
  Excellent functional neurological outcome means modified Rankin scale (mRS) scores 0-1. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Independent functional neurological outcome | Umbrella level time frame: 6 months; Substudy specific time frame may differ (details will be included in substudy-specific registration)
  Independent functional neurological outcome means modified Rankin scale (mRS) scores 0-2. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Health Related Quality of Life | Umbrella level time frame: 6 months; Substudy specific time frame may differ (details will be included in substudy-specific registration)
  Health Related Quality of Life based on EuroQol 5 Dimension 5 Level (EQ-5D-5L).The EQ-5D-5L is a generic instrument for describing and valuing health. It assesses five domains: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five response categories corresponding to: no problems, slight, moderate, severe and extreme problems.
Total length of hospital stay | Umbrella level time frame: 6 months; Substudy specific time frame may differ (details will be included in substudy-specific registration)
  Total length of hospital stay refers to the number of days from the date of hospital admission to the date of discharge.

OTHER OUTCOMES:
Mortality | Umbrella level time frame: 6 months; Substudy specific time frame may differ (details will be included in substudy-specific registration)
  Mortality status equals to death which will be collected at all visits during the trial period

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- See also: A Multicenter, RAndomlzed, coNtrolled, umBrella Trial fOr Minimally Invasive Neurosurgery With Al-assisted Robotic Guidance for Large Basal Ganglia Hemorrhage (RAINBOW-LBH) — https://clinicaltrials.gov/study/NCT06484374
- See also: A Multicenter, RAndomlzed, coNtrolled, umBrella Trial fOr Minimally Invasive Neurosurgery With Al-assisted Robotic Guidance for Moderate Basal Ganglia Hemorrhage (RAINBOW-MBH) — https://clinicaltrials.gov/study/NCT06465719
- See also: A Multicenter, RAndomlzed, coNtrolled, umBrella Trial fOr Minimally Invasive Neurosurgery With Al-assisted Robotic Guidance for IntraVentricular Hemorrhage (RAINBOW-IVH) — https://clinicaltrials.gov/study/NCT06486480
- See also: A Multicenter, RAndomlzed, coNtrolled, umBrella Trial fOr Minimally Invasive Neurosurgery With Al-assisted Robotic Guidance for BrainStem Hemorrhage (RAINBOW-BSH) — https://clinicaltrials.gov/study/NCT06459427